CLINICAL TRIAL: NCT01605890
Title: ANRS 159 VIH-2 : Trial Evaluating a First Line Combination Therapy With Raltegravir, Emtricitabine and Tenofovir in HIV-2 Infected Patients
Brief Title: Trial Evaluating a First Line Combination Therapy With Raltegravir, Emtricitabine and Tenofovir in HIV-2 Infected Patients
Acronym: VIH-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005038-20; ANRS 159 VIH-2
Record Dates: First submitted 2012-05-22; First posted 2012-05-25 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-09

CONDITIONS: HIV-2 Infection
Keywords: HIV-2
MeSH Terms: interventions — Emtricitabine; Tenofovir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- raltegravir / emtricitabine / tenofovir disoproxil fumarate (Experimental)
  Interventions: Drug: emtricitabine / tenofovir disoproxil fumarate / raltegravir .

INTERVENTIONS:
Drug: emtricitabine / tenofovir disoproxil fumarate / raltegravir . — emtricitabine : 200 mg/day and tenofovir disoproxil fumarate : 300 mg/day, included in one pill of Truvada® QD.
  raltegravir : 400 mg x 2/day, 400 mg in one pill of Isentress® BID.

SUMMARY:
The HIV-2 is less common ie 1-2 million people in West Africa. HIV-2 does have the same sensitivity to antiretroviral treatment (ART) compared to HIV-1. The ART strategies that are appropriate for the HIV-1 infection are not as effective for HIV-2. Classical triple therapy including PI is less effective for HIV-2. Also, the choice of ARTs in a second line treatment is limited. The first line optimal treatment has to be defined by a prospective and randomized evaluation of other strategies. The primary endpoint will be adapted to the specificity of the HIV-2 infection. The 1st step is to define, with a phase II clinical trial, whether a strategy including 2 NRTIs and raltegravir, as an alternative strategy to the classical triple therapy, shows an immunovirological response, at least, as good as the one obtained with the triple therapy. The hypothesis is that the low ART response observed in HIV-2 infection is due to a low virological strength of the ARTs used and that the combination of 2 NRTIs and raltegravir should show a therapeutic success of at least 50% at week 48.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* HIV-2 mono infection, confirmed by ELISA and Western Blot test or Immunoblot,
* antiretroviral treatment-naive, whatever the duration and indication of prior treatments,
* indication to treatment, with at least one of the following criteria : type B or C events, CD4 lymphocytes count below 500/mm3 at screening-visit or CD4 lymphocytes count decrease of at least 50 cell/µL/year over the last 3 years with the last CD4 lymphocytes count within -/+ 10 % of the nadir, plasma HIV-2 RNA load over or equal to 100 copies/mL at screening-visit,
* Pneumocystis prophylaxis if CD4 lymphocytes count below 200/mm3, combined to a toxoplasmosis prophylaxis in case of a positive toxoplasmosis serology,
* French residency for at least one year,
* Written informed consent, signed by the participant and the investigator (at the latest on the screening-visit and prior any study related intervention)
* Affiliate or beneficiary of a social security system (State Medical Assistance is not a social security scheme).

Exclusion Criteria:

* Absence of effective contraception method(women),
* Pregnancy, breastfeeding or wish for pregnancy during the trial,
* Curative treatment of a progressive opportunistic infection not compatible with those evaluated in the present study,
* Malignant or tumorous affection requiring chemotherapy or radiotherapy,
* Decompensated cirrhosis,
* Viral hepatitis C with a Metavir score over F2,
* Hemoglobinemia below 7g/dL, polynuclear neutrophils below 500/mm3, platelets below 50 000/mm3, creatinine clearance below 50 mL/mn, transaminase, alkaline phosphatase or bilirubin over 2.5N,
* Contraindication to one of the excipients of study treatments,
* Insuline-dependent diabetes mellitus not well controlled (with glycated haemoglobin (HbA1C) over 7%),
* Long-term corticosteroid treatment (more than 3 weeks of treatment),
* Judicial protection, legal guardianship,
* Participation in other therapeutic trial or comprising an exclusion period ongoing at the time of the screening-visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Matheron, Pr, Study Chair — Hopital Bichat-Claude Bernard
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

REFERENCES:
- [Derived] Matheron S, Descamps D, Gallien S, Besseghir A, Sellier P, Blum L, Mortier E, Charpentier C, Tubiana R, Damond F, Peytavin G, Ponscarme D, Collin F, Brun-Vezinet F, Chene G; France REcherche Nord&Sud Sida-Hiv Hepatites (ANRS) 159 HIV-2 Trial Study Group. First-line Raltegravir/Emtricitabine/Tenofovir Combination in Human Immunodeficiency Virus Type 2 (HIV-2) Infection: A Phase 2, Noncomparative Trial (ANRS 159 HIV-2). Clin Infect Dis. 2018 Sep 28;67(8):1161-1167. doi: 10.1093/cid/ciy245. PMID 29590335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled ART-naïve adults infected with HIV-2 only with history of CDC group B or C event, or a CD4 count <500 cells/μL, or a CD4 decrease >50 cells/μL/year over the past 3 years, or a confirmed plasma HIV-2 RNA (pVL) ≥100 copies (cp) /mL from 18 hospital centers in France.The last participant completed in December 2015.
Pre-assignment Details: Of the 38 participants screened between July 2012 and January 2015, 30 (78.9%) participants were finally included.
Period: Overall Study
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Started | 30
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48.8 [46.0 to 52.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Therapeutic Success
Description: The participants will be considered in therapeutic success at Week 48 if they did not present any of the following events:
  * Plasma HIV-2 RNA load over or equal to 100 copies/mL, starting from Week 24 and confirmed within the next 4 weeks,
  * CD4 lymphocytes gain below 100/mm3 at Week 48 compared to the CD4 lymphocytes counts average between Week-4 and Week 0,
  * Raltegravir permanent discontinuation,
  * Death from any cause,
  * New B or C events confirmed by an endpoint review committee
Time Frame: at Week 48
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 30
percentage of participants | 40 [22.7 to 59.4]

2. Secondary Outcome: Median Change in CD4 Lymphocytes Count at Week 12
Time Frame: between Week 0 and Week 12
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 30
cells/µL | 73 [2 to 143]

3. Secondary Outcome: Number of Clinical and Biological Events
Time Frame: from Week 0 to Week 48
Measure: Number; unit: clinical and biological events
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 30
clinical and biological events | 61

4. Secondary Outcome: Median Change of CD4 Lymphocytes at Week 48
Time Frame: between Week 0 and Week 48
Measure: Median (Inter-Quartile Range); unit: cells/µL
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 28
cells/µL | 87 [38 to 213]

5. Secondary Outcome: Percentage of Patients With Plasma HIV-2 RNA < 40 Copies/mL
Time Frame: between Week 0 and Week 48
Measure: Number; unit: percentage of participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 28
percentage of participants | 96.4

6. Secondary Outcome: Number of Participants With Clinical Progression
Description: Clinical progression is defined as the switch:
  * from category A to B, C or death.
  * from category B to C or death.
Time Frame: from Week 0 to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 30
Participants | 0

7. Secondary Outcome: Minimal Observed Percentage of Participants With Moderate to Good Adherence Evaluated With ANRS Self-administered Questionnaire of Adherence
Time Frame: from Week 4 to Week 48
Population: Number of participants with available questionnaire of adherence
Measure: Number; unit: percentage of participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 21
percentage of participants | 76

8. Secondary Outcome: Number of Virological Failure Participants With Resistance Mutations
Description: Virological failure is defined as plasma HIV-2 RNA load over or equal to 100 copies/mL after plasma HIV-2 RNA load below 100copies/mL, confirmed with a retest within the 4 following weeks. The number and type of mutations in the RT and integrase genes compared to week 0 is being reported.
Time Frame: from Week 0 to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 30
Participants | 1

9. Secondary Outcome: Number of Participants With Treatment Switch or Discontinuation
Description: Overall (regardless of the molecule)
Time Frame: from Week 0 to Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 30
Participants | 4

10. Secondary Outcome: Number of Participants With >6 Copies of HIV-2 DNA in Plasma at Week 48
Time Frame: at Week 48
Population: Participants with available measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 26
Participants | 3

11. Secondary Outcome: Minimal Median of the Lower Dimension Out of the 4 Dimensions of the Quality of Life Questionnaire
Description: The quality of life questionnaire is the Professional Quality of Life (PROQOL) questionnaire, including 4 dimensions:
  Physical health and symptoms, Relationship with others, Mental and cognitive functioning and Treatment impact For each scale, a score ranging from 0 (the worst answer) to 100 (the best answer) is calculated.
Time Frame: from Week 0 to Week 48
Population: Participants with available PROQOL questionnaire
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 22
Score on a scale | 45 [20 to 75]

12. Secondary Outcome: Number of Participants With >6 Copies of HIV-2 DNA in Plasma at Week 24
Time Frame: Week 24
Population: Participants with available measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 24
Participants | 5

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate (N=30)
Lacunar ischemic stroke (Nervous system disorders) | 1 (1) — Hospitalisation or prolongation of existing Hospitalisation
Helicobacter pylori gastritis, Escherichia coli cystitis (Infections and infestations) | 1 (1) — Also functionnal colopathy referring to the SOC=Gastrointestinal disorders
Suspected recurrence of bronchopulmonary cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hospitalisation or prolongation of existing Hospitalisation
Truvada overdose without any adverse event (Injury, poisoning and procedural complications) | 1 (1) — Other medically important condition
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir / Emtricitabine / Tenofovir Disoproxil Fumarate (N=30)
Nausea (Gastrointestinal disorders) | 5 (5)
Asthenia (General disorders) | 4 (4)
Headache (Nervous system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Backache (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Leuco-neutropenia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No